CLINICAL TRIAL: NCT05615038
Title: A Comparison of Contact Aspiration Versus Stent Retriever for Acute Basilar Artery Occlusion: A Multicentre, Prospective, Open-label, Blind Endpoint, Randomized Controlled Trial
Brief Title: A Comparison of Contact Aspiration Versus Stent Retriever for Acute Basilar Artery Occlusion
Acronym: ANGEL-COAST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Zhongrong Miao, Director of Interventional Neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2022-123-03
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-02

CONDITIONS: Basilar Artery Occlusion; Endovascular Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contact aspiration first line thrombectomy (Experimental): Patients will have the mechanical thrombectomy by first-line contact aspiration
  Interventions: Procedure: Contact aspiration Thrombectomy
- Stent retriever first line thrombectomy (Active Comparator): Patients will have the mechanical thrombectomy by first-line stent retriever
  Interventions: Procedure: Stent retriever thrombectomy

INTERVENTIONS:
Procedure: Contact aspiration Thrombectomy — Contant aspiration is an approach that utilizes the advantages of large-bore aspiration catheters that can be easily tracked and introduced into the cerebral circulation to directly remove the thrombus via negative pressure aspiration.
  Arms: Contact aspiration first line thrombectomy
Procedure: Stent retriever thrombectomy — Stent retriever thrombetomy is an approach that utilize sself-expandable stent for thrombectomy. The stent retriever is expanded to capture the thrombus, which immediately may restore blood flow.
  Arms: Stent retriever first line thrombectomy

SUMMARY:
Compare the effectiveness and safety of contact aspiration (CA) and stent retriever (SR) in acute ischemic stroke patients with basilar artery occlusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years;
2. Acute basilar artery occlusion confirmed by CTA/MRA/DSA;
3. Last known well to puncture time≤24 hours;
4. pc-ASPECTS score≥6 points;
5. Baseline NIHSS score≥10 points;
6. Consent to endovascular treatment;
7. Informed consent signed.

Clinical Exclusion Criteria:

1. Baseline mRS≥3 points;
2. Known or suspected severe basilar artery stenosis (>70%) or chronic occlusion based on history, imaging, or clinical manifestations;
3. Refractory hypertension that is difficult to be controlled by drugs (defined as persistent systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg)
4. Genetic or acquired hemorrhagic tendency, coagulation factor deficiency or on anticoagulant therapy and International Normalized Ratio (INR) > 3.0;
5. Laboratory tests: baseline blood glucose <50mg/dl (2.8mmol/L) or >400mg/dl (22.2mmol/L); Baseline platelet count <50×109/L;
6. Known severe allergy (more severe than skin rash) to contrast agents uncontrolled by medications;
7. Females who are pregnant, or those of childbearing, potential with positive urine or serum beta Human Chorionic Gonadotropin test;
8. Other circumstances that the investigator considers inappropriate for participation in the trial or that may pose significant risks to patients (such as inability to understand and/or follow the study procedures and/or follow up due to mental disorders, cognitive or emotional disorders).

Imaging Exclusion Criteria:

1. CT or MR evidence of acute intracranial hemorrhage (the presence of microbleeds on MRI is allowed);
2. Midline shift or herniation, mass effect with effacement of the ventricles;
3. Complete cerebellar infarct on CT or MRI with significant mass effect and compression of the 4-th ventricle;
4. Complete bilateral thalamic infarction on CT or MRI;
5. Inability to endovascular treatment due to Excessive tortuosity, variation, or dissection of the artery;
6. Subjects with occlusions in both intracranial vertebral arteries;
7. Subjects with occlusions in both anterior and posterior circulation;
8. Evidence of intracranial tumor (except small meningioma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of first pass effect (FPE) | 24 hours
  [The definition of FPE: 1) single pass/use of the device; 2)recanalization of the large vessel occlusion to eTICI 2C/3;3) no use of rescue therapy.]

SECONDARY OUTCOMES:
Rate of complete reperfusion (eTICI 3) after first-line thrombectomy strategy and at the end of endovascular procedure | 24 hours
  eTICI： grade 0: no perfusion noted (0% reperfusion) grade 1: reduction in thrombus but without any resultant filling of distal arterial branches grade 2 grade 2a: reperfusion of 1-49% of the territory grade 2b50: reperfusion of 50-66% of the territory grade 2b67: reperfusion of 67-89% of the territory grade 2c: extensive reperfusion of 90-99% of the territory grade 3: complete or full reperfusion (100% reperfusion)
Rate of near to complete reperfusion (eTICI 2c/3) after first-line thrombectomy strategy and at the end of endovascular procedure | 24 hours
  eTICI： grade 0: no perfusion noted (0% reperfusion) grade 1: reduction in thrombus but without any resultant filling of distal arterial branches grade 2 grade 2a: reperfusion of 1-49% of the territory grade 2b50: reperfusion of 50-66% of the territory grade 2b67: reperfusion of 67-89% of the territory grade 2c: extensive reperfusion of 90-99% of the territory grade 3: complete or full reperfusion (100% reperfusion)
Rate of successful reperfusion (eTICI 2b/2c/3) after first-line thrombectomy strategy and at the end of endovascular procedure | 24 hours
  eTICI： grade 0: no perfusion noted (0% reperfusion) grade 1: reduction in thrombus but without any resultant filling of distal arterial branches grade 2 grade 2a: reperfusion of 1-49% of the territory grade 2b50: reperfusion of 50-66% of the territory grade 2b67: reperfusion of 67-89% of the territory grade 2c: extensive reperfusion of 90-99% of the territory grade 3: complete or full reperfusion (100% reperfusion)
Rate of Arterial Occlusive Lesion (AOL) recanalization score 3 after first-line thrombectomy strategy and at the end of endovascular procedure | 24 hours
  AOL recanalization score is evaluated between 0 to 3:
  0 indicates no recanalization of the primary occlusive lesion;
  1. indicates incomplete or partial recanalization of the primary occlusive lesion with no distal flow;
  2. indicates incomplete or partial recanalization of the primary occlusive lesion with any distal flow;
  3. indicates complete recanalization of the primary occlusive with any distal flow.
Groin puncture time to successful reperfusion time (min) | 24 hours
  evaluated in minutes
The difference of NIHSS score between 24-hour and baseline | 24 hours
  NIHSS (National Institutes of Health Stroke Scale) score is evaluated between 0-42 0 is normal and 42 maximal gravity
Modified Rankin Score (mRS) at 90±14 days (shift analysis) | 90 days
  mRS is evaluated between 0 to 6. A score of 0 indicates that there is no disability and a score of 6 indicates death.
Rate of mRS 0-1 at at 90±14 days | 90 days
  mRS is evaluated between 0 to 6. A score of 0 indicates that there is no disability and a score of 6 indicates death.
Rate of mRS 0-2 at at 90±14 days | 90 days
  mRS is evaluated between 0 to 6. A score of 0 indicates that there is no disability and a score of 6 indicates death.
Rate of mRS 0-3 at at 90±14 days | 90 days
  mRS is evaluated between 0 to 6. A score of 0 indicates that there is no disability and a score of 6 indicates death.
Quality of life at 90±14 days assessed by EuroQol 5D-5L scale | 90 days
  EuroQol 5D-5L comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions.
  This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Rate of symptomatic intracranial hemorrhage within 48 hours (according to Heidelberg Bleeding Classification) | 48 hours
  Heidelberg Bleeding Classification:
  1. Hemorrhagic transformation of infarcted brain tissue 1a HI1 Scattered small petechiae, no mass effect 1b HI2 Confluent petechiae, no mass effect 1c PH1 Hematoma within infarcted tissue, occupying <30%, no substantive mass effect 2 Intracerebral hemorrhage within and beyond infarcted brain tissue PH2 Hematoma occupying 30% or more of the infarcted tissue, with obvious mass effect 3 Intracerebral hemorrhage outside the infarcted brain tissue or intracranial-extracerebral hemorrhage 3a Parenchymal hematoma remote from infarcted brain tissue 3b Intraventricular hemorrhage 3c Subarachnoid hemorrhage 3d Subdural hemorrhage
Rate of any intracranial hemorrhage within 48 hours (according to Heidelberg Bleeding Classification) | 48 hours
  Heidelberg Bleeding Classification:
  1. Hemorrhagic transformation of infarcted brain tissue 1a HI1 Scattered small petechiae, no mass effect 1b HI2 Confluent petechiae, no mass effect 1c PH1 Hematoma within infarcted tissue, occupying <30%, no substantive mass effect 2 Intracerebral hemorrhage within and beyond infarcted brain tissue PH2 Hematoma occupying 30% or more of the infarcted tissue, with obvious mass effect 3 Intracerebral hemorrhage outside the infarcted brain tissue or intracranial-extracerebral hemorrhage 3a Parenchymal hematoma remote from infarcted brain tissue 3b Intraventricular hemorrhage 3c Subarachnoid hemorrhage 3d Subdural hemorrhage
Rate of procedure-related complications, included arterial dissection, embolization in a new territory, arterial perforation and subarachnoid haemorrhage | 24 hours
All cause of mortality at 90±14 days | 90 days

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Anzhen Hospital, Beijing, Beijing Municipality
  - Beijing Daxing District People's Hospital, Beijing, Beijing Municipality
  - Anyang People's Hospital, Anyang, Henan
  - Zhangzhou Municipal Hospital, Zhangzhou, Henan
  - Baotou Center Hospital, Baotou, Neimenggu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Xuan S, Yang M, Sun D, Song L, Gao F, Mo D, Ma N, Pan Y, Liu L, Zhao X, Wang Y, Wang Y, Nogueira R, Miao Z. Contact aspiration versus stent retriever thrombectomy for acute basilar artery occlusion (ANGEL-COAST): rationale and design of a multicentre, prospective, randomised, open-label, blinded-endpoint trial. Stroke Vasc Neurol. 2025 Oct 28:svn-2025-004232. doi: 10.1136/svn-2025-004232. Online ahead of print. PMID 41151802